CLINICAL TRIAL: NCT04190303
Title: NIHR Global Health Research Group on Brain Infections Study: Establishing a Standard Care Package to Improve Diagnosis and Early Hospital Management of Patients With Suspected Acute Brain Infections in Low and Middle Income Countries
Brief Title: BIGlobal Intervention Study: Improving Diagnosis and Management of Suspected Brain Infections Globally
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Christian Medical College, Vellore, India (Other); National Institute of Mental Health and Neuro Sciences, India (Other); Oswaldo Cruz Foundation (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Kamuzu University of Health Sciences (Other); University of Warwick (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Principal Investigator, Tom Solomon, Professor, University of Liverpool
Other Study IDs: UoL001430 - 4069
Record Dates: First submitted 2019-12-01; First posted 2019-12-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Meningitis; Encephalitis; Abscess Brain
MeSH Terms: conditions — Meningitis; Encephalitis; Brain Abscess

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline (pre-intervention): Current routine care
- Post-intervention: Care following development and delivery of the system-level intervention
  Interventions: Other: Pragmatic, multi-component package

INTERVENTIONS:
Other: Pragmatic, multi-component package — This system-level intervention will be tailored to the needs and capacity of each hospital site, co-developed with policymakers and hospital staff
  Groups: Post-intervention

SUMMARY:
Background: Patients with suspected brain infections pose major challenges to low and middle income countries, including their disproportionately high burden, diverse causes with inadequate surveillance, requirement for invasive and expensive tests, and the difficulty of management without a clear diagnosis. This is all compounded by resource and system constraints. Few studies have attempted to improve the care of these people in resource-limited settings.

Aim: This study sets out to improve the diagnosis and early management of people with suspected acute (<28 days of symptoms) brain infections in low and middle income countries, using a coordinated thematic approach.

Outcomes: The primary outcome will be proportion of people with suspected acute brain infection receiving a diagnosis. Secondary outcomes will include mortality, length of stay in hospital, quality of life, degree of disability, and proportion having a lumbar puncture test.

Participants: Children and adults with features consistent with an acute brain infection, including meningitis and encephalitis, will be recruited at a variety of hospitals in Brazil, India and Malawi.

Study procedures: An assessment of current practice and capabilities at each hospital, including patient and sample journey observations and interviews with healthcare staff, will identify barriers to optimal care. Using this, a sustainable pragmatic multi-component intervention will be produced, with components modifiable to each hospital's needs. Outcomes will be reassessed post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, infants and children presenting to a study hospital with symptoms and/or signs suggestive of acute brain infection, which could be suspected encephalitis, suspected meningitis, or alternative features raising suspicion of brain infection.
2. Symptom duration of less than 4 weeks.

Exclusion Criteria:

1. Neonates, i.e. children under the age of 28 days.
2. People with pre-existing indwelling ventricular devices (e.g. extra-ventricular drains, ventriculo-peritoneal shunts) or other implants in contact with the meninges or brain (e.g. deep brain stimulators).
3. People without an indwelling device, having undergone neurosurgical procedures within the preceding 12 months.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to a study hospital with symptoms and/or signs suggestive of an acute brain infection.
Sampling Method: Probability Sample
Enrollment: 2233 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Microbiological diagnosis | During hospital admission, or at 30 days if participant still in hospital
  Proportion of patients achieving microbiological diagnosis
Syndromic diagnosis | During hospital admission, or at 30 days if participant still in hospital
  Proportion of patients achieving syndromic diagnosis

SECONDARY OUTCOMES:
Proportion receiving, and time to lumbar puncture | During hospital admission, or at 30 days if participant still in hospital
  Proportion of study participants receiving a lumbar puncture, and time to lumbar puncture
Proportion having appropriate cerebrospinal fluid investigations | During hospital admission, or at 30 days if participant still in hospital
  All of: cell count, total and differential; CSF protein concentration; CSF glucose concentration; paired serum/blood glucose concentration; microscopy and culture for bacteria
Mortality | At 30 days
  All-cause
Length of stay in hospital | During hospital admission, or at 30 days if participant still in hospital
  Duration of hospital admission
Time to appropriate empirical therapy | During hospital admission, or at 30 days if participant still in hospital
  Time to appropriate empirical anti-infective therapy
Time to appropriate definitive therapy | During hospital admission, or at 30 days if participant still in hospital
  Time to appropriate definitive anti-infective therapy
Quality of life score | At hospital discharge, or at 30 days if participant still in hospital
  Using EuroQol EQ-5D questionnaires scoring 5 domains at levels 1-3 each, and an overall health state from 0 to 100.
Quality of life score | At 30 days after presentation to hospital
  Using EuroQol EQ-5D questionnaires scoring 5 domains at levels 1-3 each, and an overall health state from 0 to 100.
Liverpool Outcome Score | At hospital discharge, or at 30 days if participant still in hospital
  Score measuring neurological function after brain infection, reporting a lowest score of 15 domains between 2 and 5, and a total score with range 33-75.
Liverpool Outcome Score | At 30 days after presentation to hospital
  Score measuring neurological function after brain infection, reporting a lowest score of 15 domains between 2 and 5, and a total score with range 33-75.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Solomon, PhD, Principal Investigator — Institute of Infection & Global Health, University of Liverpool
Locations (4):
- FioCruz, Recife, Brazil
- India (2):
  - National Institute of Mental Health and Neurosciences, Bangalore
  - Christian Medical College, Vellore
- Malawi Liverpool Wellcome Trust, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh B, Lipunga GD, Thangavelu P, Dhar S, Ferreira Cronemberger L, Abhilash KPP, Abraham AM, de Brito CAA, Brito Ferreira ML, Chandrashekar N, Duarte R, Fajardo Modol A, Ghale BC, Kang G, Gowda VK, Kuriakose K, Lant S, Mallewa M, Mbale E, Moore SC, Mwangalika G, Kamath PBT, Navvuga P, Nyondo-Mipando AL, Phiri TJ, Pimentel Lopes de Melo C, Pradeep BS, Rawlinson R, Sheha I, Thomas PT, Newton CR, de Sequeira PC, Sejvar JJ, Dua T, Turtle L, Verghese VP, Arraes LWMS, Desmond N, Easton A, Jones JA, Lilford RJ, Netravathi M, McGill F, Michael BD, Mwapasa V, Griffiths MJ, Parry CM, Ravi V, Burnside G; Brain Infections Global Intervention Study Group; Cornick J, Franca RFO, Desai AS, Rupali P, Solomon T. A multifaceted intervention to improve diagnosis and early management of hospitalised patients with suspected acute brain infections in Brazil, India, and Malawi: an international multicentre intervention study. Lancet. 2025 Mar 22;405(10483):991-1003. doi: 10.1016/S0140-6736(25)00263-6. Epub 2025 Mar 10. PMID 40081400